CLINICAL TRIAL: NCT01836289
Title: High-dose Cyclophosphamide for Severe Refractory Crohn Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Too difficult to recruit given new Crohn's medications approved
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00052668
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Crohn's Disease; Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High-dose Cyclophosphamide (Experimental): High-dose Cyclophosphamide
  Interventions: Drug: High-dose Cyclophosphamide

INTERVENTIONS:
Drug: High-dose Cyclophosphamide
  Other Names: Endoxan®; Cytoxan®; CTX; Neosar®; Procytox®; Revimmune™

SUMMARY:
This research is being done to see if people with Crohn's disease who receive high-dose cyclophosphamide have an improvement of their disease, how long the benefit may last, and how safe cyclophosphamide is. This study is for patient with medically refractory disease that is not easily amenable to surgery.

Cyclophosphamide is an FDA-approved chemotherapy medication that is also frequently used to treat autoimmune illness; use of cyclophosphamide for autoimmune disease is not approved by the FDA. An autoimmune illness is when the immune system mistakenly attacks self, targeting the cells, tissues, and organs of a person's own body. There are many different autoimmune diseases and they can each affect the body is different ways. Crohn's disease is an autoimmune disease that primarily affects the small and large intestines. High dose-cyclophosphamide has been successfully used to treat Crohn's, primarily as part of a conditioning regimen for autologous stem cell transplantation. However, this therapy is limited in Crohn's because of it's serious infectious risks. This current study involves using high-dose cyclophosphamide without need for stem cell transplantation. This appears to be a safer approach in other autoimmune illnesses that have been studied.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age, males and females will be eligible
* Moderate to severe Crohn's Disease (CD) with CDAI > 220, in addition to evidence of ulceration on ileocolonoscopy or active disease on small bowel imaging (in patients with an ostomy, CDAI criteria do not apply)
* Disease progression (primary or secondary non-responder, or reaction to) to at least one anti-tumor necrosis factor (TNF) agent (infliximab, adalimumab, certolizumab pegol), and additionally had disease progression despite one of the following immunosuppressant drugs: azathioprine, 6-mercaptopurine, methotrexate, cyclosporine, natalizumab, vedolizumab
* Willingness to participate in a clinical trial
* Approval by Enrollment Panel, who will collectively decide on the appropriateness of possible study study participants

Exclusion Criteria:

* Pregnant or nursing women
* Sexually active men and women who do not agree to use effective means of birth control during treatment period
* Evidence of primarily fibrostenosing disease without active inflammatory disease on disease staging
* Co-morbid conditions including cardiac disease with an ejection fraction of < 45%, chronic renal failure with serum creatinine > 2.0, liver disease with total bilirubin > 2.0, (excluding hyperbilirubinemia secondary to Gilbert's disease) or transaminitis > 3x upper limit of normal.
* History of serious allergic reaction to cyclophosphamide
* History of malignancy in the last 5 years (excluding non-melanomatous skin cancers)
* Patients who are pre-terminal
* Toxic megacolon
* Active infection
* White blood cell count < 3000 cells/ul, platelets < 100K / ul, hemoglobin < 10.0 g/dL
* Any use of thiopurines, methotrexate or anti-TNF agents in the previous four weeks prior to treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety of the High-Dose Cyclophosphamide (HDC) protocol | 3 Years
  Tablulation of serious adverse events associate with the HDC protocol

SECONDARY OUTCOMES:
HDC-Induced Steroid-free remission | 3 Years
  To determine if HDC therapy can induce and maintain a steroid-free clinical remission (defined as CDAI<150) at 12 and 52 weeks. Applies to patients without an existing ostomy.
HDC-Induced Mucosal Healing | 3 Years
  To determine if HDC therapy can induce sustained mucosal healing defined as absence of ulcers on colonoscopy
Improvement in patient reported quality of life | 3 years
  To determine if HDC can lead to improvement in inflammatory bowel disease questionnaire scores at weeks 12 and 52
Molecular Mechanisms of High-dose Cyclophosphamide (HiCy) Therapy | 3 Years
  To investigate the molecular mechanisms by which HiCy therapy works by analyzing the effects of HiCy on the levels of serum cytokines (using multiplex ELISA), and correlate the data with clinical activity and treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Mark G. Lazarev, MD, Principal Investigator — Johns Hopkins University